CLINICAL TRIAL: NCT03169699
Title: Acoustic Analytic Apps for Smart Telehealth Screening - Creating a Big Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore University of Technology and Design (Unknown)
Responsible Party: Sponsor
Other Study IDs: KKWCH 2016/2416
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: URTI; Cough; Cough Variant Asthma; Cough; Bronchial, With Grippe or Influenza
MeSH Terms: conditions — Cough; Cough-Variant Asthma; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cough Arm: Children age 16 years old and below with cough at presentation - Patients presenting with active or chronic or residual cough
- Well Arm: Children age 16 years old and below and Well with no presentation of cough

SUMMARY:
To develop and validate a library of cough spectrum from a target of 1000 cough acoustics. Coughs arising from upper respiratory infection, lower chest infections, asthma, allergic conditions are included in the study. Cough acoustic in absence of respiratory disease is also included.

This is a prospective observation cohort study recruiting children below the age of 16 years old in 2 arms : (1) Patients with respiratory conditions presenting with cough and (2) Well patients without active coughing.

DETAILED DESCRIPTION:
Cough is a common presentation in childhood. It is one of the early symptom of respiratory disease such as upper respiratory tract infection, cough variant asthma, allergic rhinitis, bronchitis and pneumonia. These conditions are common ailments in childhood. The history of cough and description of cough given by caretakers and patients are often vague and assessment of cough quality is often subjective. The quality of cough is often assigned a dichotomous category of dry cough and wet cough.

Computer assisted cough analysis has been developed in recent years to aid subjective classification of cough. The sound spectrum and frequencies of cough is being researched to better define the quality of cough. The quality of cough gives meaningful information about the state of the respiratory status. Cough sound analysis has been shown to rapidly diagnose pneumonia in humans using cough sound analysis and in differentiating wet and dry cough.

The investigators hypothesize that each respiratory pathology will have its spectral cough characteristics. Analysis of cough spectrum and comparing to a library of cough spectra data will be able to aid differentiation of the underlying conditions for the various cough spectrum and hence facilitating management.

The study aim is to develop a computer processing technique of cough sounds and determine their spectral characteristics for the common causes of cough to derive an assisted assay of cough spectrum for an objective assessment of cough.

ELIGIBILITY:
Inclusion Criteria:

* Cough arm 1.Children age 16 years old and below with cough at presentation- Patients presenting with active or chronic or residual cough

Well arm

1.Children age 16 years old and below and Well with no cough presentation.

Exclusion Criteria:

1. Children with severe behavioral
2. Droplet isloated cases as determined by protocol of hospital

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is a prospective observation cohort study will recruit children below the age of 16 years old.
  There will be 2 arms : (1) Patients with respiratory conditions presenting with cough and (2) well patient without cough.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute phase acoustic spectrum Analysis | Day 0-7
  Acoustic classifiers

SECONDARY OUTCOMES:
Recovery or Chronic phase acoustic spectrum analysis | Day 7-30
  Acoustic classifiers

CONTACTS AND LOCATIONS:
Overall Officials: Hwan Ing Hee, MBBCH BAO, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KKWCH, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] B T B, Hee HI, Teoh OH, Lee KP, Kapoor S, Herremans D, Chen JM. Asthmatic versus healthy child classification based on cough and vocalised /a:/ sounds. J Acoust Soc Am. 2020 Sep;148(3):EL253. doi: 10.1121/10.0001933. PMID 33003873